CLINICAL TRIAL: NCT01014546
Title: A Phase I Study of Oral Arsenic Trioxide With or Without Ascorbic Acid in Adults With Myelofibrosis
Brief Title: Arsenic Trioxide With or Without Ascorbic Acid in Treating Patients With Myelofibrosis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: low accrual
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: Cephalon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 154609; NCI-2009-01660 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 154609 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2009-11-16; First posted 2009-11-17 (Estimated); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Essential Thrombocythemia; Polycythemia Vera; Primary Myelofibrosis
MeSH Terms: conditions — Thrombocythemia, Essential; Polycythemia Vera; Primary Myelofibrosis | interventions — Arsenic Trioxide; arsenous acid; Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (arsenic trioxide with or without ascorbic acid) (Experimental): Patients receive arsenic trioxide PO QD in orange juice on days 1-21. Patients may also receive ascorbic acid PO QD on days 1-21. Treatment repeats every 28 days for up to 168 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Arsenic Trioxide; Dietary Supplement: Ascorbic Acid; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study

INTERVENTIONS:
Drug: Arsenic Trioxide — Given PO
  Other Names: Arsenic (III) Oxide; Arsenic Sesquioxide; Arsenous Acid; Arsenous Acid Anhydride; Arsenous Oxide; Trisenox; White Arsenic
Dietary Supplement: Ascorbic Acid — Given PO
  Other Names: 2-(1,2-dihydroxyethyl)-4,5-dihydroxy-furan-3-one; Asorbicap; C Vitamin; C-Long; Ce-Vi-Sol; Cecon; Cenolate; Cetane; Cevalin; L-Ascorbic Acid; VIT C; Vitamin C; Vitamin-C
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of arsenic trioxide with or without ascorbic acid in treating patients with myelofibrosis. Drugs used in chemotherapy, such as arsenic trioxide, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving arsenic acid together with ascorbic acid may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and maximum tolerated dose of oral arsenic trioxide with or without ascorbic acid in subjects with myelofibrosis.

SECONDARY OBJECTIVES:

I. To estimate the incidence, severity, and attribution of treatment-emergent adverse events.

II. To estimate the rate of complete or major clinical-hematological response from treatment with arsenic trioxide and ascorbic acid in this subject population as measured by the International Working Group for Myelofibrosis Research and Treatment (IWG-MRT) response criteria.

III. To measure arsenic trioxide levels in the plasma of patients treated with and without ascorbic acid on this protocol.

IV. To estimate the efficacy of arsenic trioxide with ascorbic acid in subjects with myelofibrosis, as determined by a reduction in Janus kinase 2 (JAK2) V617F, JAK22T875N, and mutations of the thrombopoietin receptor (MPL515L/K) allele frequency in peripheral blood neutrophils.

V. To examine the effect of treatment on biological markers of myeloproliferation, cytokine production and hematopoietic stem cell mobilization. In particular, the following markers of disease will be measured: cluster of differentiation (CD)34+ cell count in peripheral blood measured by cytofluorimetry, plasma vascular endothelial growth factor (VEGF), transforming growth factor-beta (TGF-B), stromal cell-derived factor-1 (SDF-1), neutrophil elastase levels by commercial assays.

VI. To examine single nucleotide polymorphism (SNP) in the arsenic trioxide pathway in subjects with myelofibrosis treated with arsenic trioxide and ascorbic acid.

OUTLINE: This is a dose-escalation study of arsenic trioxide.

Patients receive arsenic trioxide orally (PO) once daily (QD) in orange juice on days 1-21. Patients may also receive ascorbic acid PO QD on days 1-21. Treatment repeats every 28 days for up to 168 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 4 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary myelofibrosis, essential thrombocythemia related myelofibrosis, or polycythemia vera related myelofibrosis requiring therapy, including:

  * Those previously treated and relapsed or refractory
  * Or, if newly diagnosed, with intermediate or high risk according to Lille scoring system (adverse prognostic factors are: hemoglobin [Hb] < 10 g/dl, white blood cell count [WBC] < 4 or > 30 x 10^9/L; risk group: 0 = low, 1 = intermediate, 2 = high)
  * Or with symptomatic splenomegaly (must be >= 23 cm by ultrasound in the longitudinal axis)
* Signed informed consent: patients must have signed consents for both the arsenic trioxide with ascorbic acid protocol and for the hematologic malignancy procurement protocol to be eligible to participate
* Patients must have been off any primary myelofibrosis (PMF)-directed experimental therapy for 4 weeks prior to entering this study and have recovered from the toxic effects (grade 0-1) of that therapy; treatment with hydroxyurea and erythropoietin are permitted until study initiation
* Serum bilirubin levels =< 2 times the upper limit of the normal range for the laboratory (ULN); higher levels are acceptable if these can be attributed by treating physician to active hemolysis or ineffective erythropoiesis due to myelofibrosis
* Serum glutamic-pyruvic transaminase (SGPT) (alanine aminotransferase [ALT]) levels =< 2 x ULN
* Serum creatinine levels =< 1.5 x ULN
* Women of childbearing potential must have a negative serum or urine pregnancy test prior to arsenic trioxide treatment and should be advised to avoid becoming pregnant
* Men must be advised to not father a child while receiving treatment with arsenic trioxide
* Both women of childbearing potential and men must practice effective methods of contraception (those generally accepted as standard of care measures)
* Women of childbearing potential are women who are not menopausal for 12 months or who have not undergone previous surgical sterilization
* If the subject is a woman of childbearing potential, she must use a medically acceptable form of contraception during the study period and for 30 days thereafter
* If the subject is a man he must be surgically sterile or must use a medically approved method of contraception for the duration of the study and for 60 days following the last dose of arsenic trioxide

Exclusion Criteria:

* Nursing and pregnant females; should a woman become pregnant or suspects she is pregnant while participating in this study, she should inform her treating physician immediately
* New York Heart Association (NYHA) grade II or greater congestive heart failure
* Unstable angina
* Corrected QT interval (QTc) > 450 in the presence of potassium >= 4 mEq/L and magnesium >= 1.7 mEq/L
* Eastern Cooperative Oncology Group (ECOG) > 2
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days, or anticipation of the need for major surgical procedure during the course of the study
* Biopsy or other minor surgical procedure, excluding placement of a vascular access device or bone marrow biopsy, within 7 days prior to study enrollment
* Ongoing serious, non-healing wound, ulcer, or bone fracture
* Known hypersensitivity to any component of arsenic trioxide

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-04; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Adverse events, and their attribution throughout the study | Up to 30 days post-treatment
  The frequency of toxicities will be tabulated by grade across all dose levels and courses. The frequency of toxicities will also be tabulated for the dose chosen as the MTD.
Dose-limiting toxicity (DLT) as assessed by the National Cancer Institute (NCI) Common Toxicity Criteria (CTC) version 3.0 (Stage 1) | At 28 days
  DLT is defined as any non-hematologic treatment-emergent grade 3 or greater adverse event deemed possibly, probably, or definitely related to the study drug. Exceptions are grade 3 nausea or vomiting, unless in the setting of maximal antiemetic treatment. Hematologic toxicities are not included in the definition of a DLT. The frequency of toxicities will be tabulated by grade across all dose levels and cycles.
Maximum tolerated dose (MTD), defined as the dose level at which 0 or 1 of 6 subjects experience DLT, and 2 of 3 or 2 of 6 experience DLT at the next higher dose level, assessed by the NCI CTC version 3.0 (Stage 1) | At 28 days
  The frequency of toxicities will be tabulated by grade across all dose levels and cycles. The frequency of toxicities will also be tabulated for the dose chosen as the MTD.

SECONDARY OUTCOMES:
Change in absolute number of circulating CD34+ cells in the peripheral blood (Stage 2 only) | Baseline to 24 weeks
Change in JAK2/MPL (Stage 2 only) | Baseline to 24 weeks
Change in plasma levels of chemokines as measured by ELISA (Stage 2) | Baseline to 24 weeks
  Including: sVCAM-1, NE, MMP-2, MMP-9, SDF-1, TGF-B, and VEGF.
Change in plasma levels of cytokines as measured by ELISA (Stage 2) | Baseline to 24 weeks
  Including: sVCAM-1, NE, MMP-2, MMP-9, SDF-1, TGF-B, and VEGF.
Change in plasma levels of proteases as measured by enzyme-linked immunosorbent assay (ELISA) (Stage 2) | Baseline to 24 weeks
  Including: soluble vascular cell adhesion molecule 1 (sVCAM-1), neutrophil elastase (NE), matrix metalloproteinases 2 and 9 (MMP-2 and MMP-9), stromal cell derived growth factor-1 (SDF-1), TGF-B, and VEGF.
Disease response assessed using the IWG-MRT response criteria | Up to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Eunice Wang, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States